CLINICAL TRIAL: NCT04072029
Title: Escala de Riesgo de descompensación Corneal en cirugía de Catarata en Pacientes Con Distrofia Corneal de Fuchs
Brief Title: Risk Assessment for Progression to DMEK Following Cataract Surgery in Fuchs Endothelial Corneal Dystrophy
Status: Completed | Type: Observational
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Sponsor
Other Study IDs: 252/17
Record Dates: First submitted 2019-04-22; First posted 2019-08-28 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2019-04

CONDITIONS: Fuchs' Endothelial Dystrophy; Cataract
MeSH Terms: conditions — Fuchs' Endothelial Dystrophy; Cataract | interventions — Phacoemulsification; Lens Implantation, Intraocular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cataract - FECD: Eyes with FECD undergoing cataract surgery
  Interventions: Procedure: Phacoemulsification with intraocular lens implantation

INTERVENTIONS:
Procedure: Phacoemulsification with intraocular lens implantation — Phacoemulsification (2.2mm coaxial, viscoelastic shield, experienced surgeon) with intraocular lens implantation (acrylic hidrophobic)

SUMMARY:
Justification. Fuchs' corneal endothelial dystrophy (FECD) is one of the main causes of corneal transplantation. In many cases, the corneal decompensation derived from this dystrophy is triggered as a consequence of cataract surgery, so the dilemma of facing isolated cataract surgery or combined with endothelial keratoplasty is often raised.

Objective. The present study aims to evaluate and select the most important predictive factors for corneal decompensation after cataract surgery in patients with FECD.

Method. Prospective observational study of the preoperative and intraoperative variables presumably associated with postoperative corneal edema requiring Descemet stripping endothelial keratoplasty (DMEK). Consecutive candidates for cataract surgery with FECD will be selected and anterior segment imaging will be performed, along with a complete ophthalmological examination. Clinical, pachymetric, tmographic, densitometric, specular microscopy, and intraoperative variables will be registered.

ELIGIBILITY:
Inclusion Criteria:

* FECD grade 2 or worse (modified Krachmer scale)
* Cataract requiring surgery
* Epithelial corneal edema evident in slit lamp examination

Exclusion Criteria:

* Concurrent anterior corneal dystrophy
* History of ocular trauma, ocular surgery, previous ocular inflammation or infection,uncotroled glaucoma, amblyopia, neovascular age-related macular degeneration, or active vacular retinal disease.
* Non-collaborative or unable to receive postoperative care at our institution.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients referred for cataract surgery to the Cornea Department
Sampling Method: Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Rate of progression to endothelial keratoplasty (DMEK) | 2 months after cataract surgery
  Evaluation of baseline parameters that could predict the need for DMEK taking into account best espetacle corrected visual acuity and visual symptoms attributable to FECD and corneal edema (worse vision in the mornings, starburst or halos at night or subjective impairment of vision interfering with daily routine activities such as reading printed paper, looking at screens or driving)

SECONDARY OUTCOMES:
Best spectacle corrected visual acuity | 2 months after cataract surgery
  Measured in logMAR scale
Corneal tomography changes | 2 months after cataract surgery
  Changes in pachymetric parameters (corneal thickness at the apex, center of the pupil, thinnest point and relative pachymetry) and densitometry (central corneal light backscatter) measured by Pentacam Scheimpflug tomograpy.
Postoperative refraction | 2 months after cataract surgery and after DMEK surgery
  Postoperative subjective refraction (sphere, cylinder, axis)

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Arnalich Montiel, MD,PhD, Principal Investigator — H.U. Ramón y Cajal
Locations (1):
- Hospital Universitario Ramón y Cajal, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No